CLINICAL TRIAL: NCT00082667
Title: EGFR Pathway Modulation In Patients With Ductal Carcinoma In Situ Of The Breast
Brief Title: Gefitinib Followed By Surgery in Treating Women With Ductal Carcinoma In Situ of the Breast
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left VICC
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VICC BRE 0249; P30CA068485 (NIH); VICC-BRE-0249
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: breast cancer in situ; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Gefitinib; Surgical Procedures, Operative; Mastectomy, Segmental

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gefitinib
  Other Names: ZD 1839, Iressa
Procedure: Surgery
  Other Names: lumpectomy or mastectomy of the breast

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. It is not yet known whether surgery is more effective with or without gefitinib in treating ductal carcinoma in situ.

PURPOSE: This randomized phase II trial is studying how well gefitinib together with surgery works compared to surgery alone for the treatment of women with ductal carcinoma in situ of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare epidermal growth factor receptor (EGFR) pathway biomarker modulation in tissue samples of women with ductal carcinoma in situ (DCIS) of the breast treated with gefitinib vs placebo followed by local surgery.
* Compare the effect of these regimens on cell turnover in vivo in EGFR-positive vs EGFR-negative patients.

Secondary

* Compare the efficacy of these regimens in estrogen-receptor (ER)-positive vs ER-negative and in HER2-positive vs HER2-negative patients with DCIS.
* Correlate levels of HER2 extracellular domain with biomarker modulation in patients treated with these regimens.

OUTLINE: This is a randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral gefitinib once daily for 7-14 days or until the day before local surgery. Patients then undergo lumpectomy or mastectomy.
* Arm II: Patients receive oral placebo once daily for 7-14 days or until the day before local surgery. Patients then undergo local surgery as in arm I.

PROJECTED ACCRUAL: A total of 78 patients (39 per treatment arm) will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ (DCIS) of the breast OR mammogram highly suspicious for DCIS

  * No invasive disease
  * Not completely excised
* Epidermal growth factor receptor (EGFR) positive (> 10% of cells stained)
* Planned lumpectomy or mastectomy within the next 2-4 weeks
* Hormone receptor status:

  * Estrogen receptor status known

PATIENT CHARACTERISTICS:

Age

* 35 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 1.5 mg/dL
* SGOT ≤ 2 times upper limit of normal (ULN)
* SGPT < 1.5 times ULN
* PT and PTT ≤ 1.5 times ULN
* INR ≤ 1.5 times ULN

Renal

* Creatinine < 1.5 mg/dL

Cardiovascular

* No New York Heart Association class I-IV heart disease

Pulmonary

* No acute asthma

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Random blood sugar < 2.5 times ULN
* No known hypersensitivity to study drug or its excipients
* No nonhealing wound or fracture
* No active infection
* No other malignancy within the past 5 years except basal cell carcinoma, breast carcinoma, or carcinoma in situ of the cervix
* No psychosis or severe depression
* No other concurrent uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior trastuzumab (Herceptin®)

Chemotherapy

* At least 1 year since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* At least 1 year since prior aromatase inhibitors
* At least 1 year since prior antiestrogens or luteinizing hormone-releasing hormone agonists or antagonists
* No concurrent glucocorticoids
* Concurrent oral contraceptives allowed
* Concurrent hormone replacement therapy allowed

Radiotherapy

* At least 1 year since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior oncologic or other major surgery
* No prior organ allograft

Other

* Recovered from all prior therapy (except alopecia)
* More than 30 days since prior non-approved or investigational drugs
* No prior definitive local therapy
* No prior immunosuppressive therapy
* No prior gefitinib
* No other prior EGFR inhibitors
* No other concurrent cytotoxic drugs
* No concurrent warfarin for anticoagulation
* No concurrent CYP3A4 inducers, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
  * Ethosuximide
  * Griseofulvin
  * Nafcillin
  * Nelfinavir
  * Nevirapine
  * Oxcarbazepine
  * Phenylbutazone
  * Primidone
  * Rifabutin
  * Rofecoxib
  * Sulfamethazine
  * Sulfinpyrazone
  * Troglitazone
* No concurrent antiretroviral treatment for HIV-positive patients

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2002-10; Primary Completion 2004-07 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Compare epidermal growth factor receptor (EGFR) pathway biomarker modulation in tissue samples of women with ductal carcinoma in situ (DCIS) of the breast treated with gefitinib vs placebo followed by surgery. | at time of surgery, after 7-14 days of gefitinib

SECONDARY OUTCOMES:
Compare the effect of gefitinib vs. placebo, followed by surgery on cell turnover in vivo in EGFR-positive vs. EGFR-negative patients | at time of surgery, after 7-14 days of gefitinib
Compare the effects of gefitinib in ER-positive vs. ER-negative DCIS and in HER2-positive vs. HER2-negative DCIS | at time of surgery, after 7-14 days of gefitinib

OTHER OUTCOMES:
Correlate levels of HER2 extracellular domain in ER-positive vs. ER-negative and in HER2-positive cs. HER2-negative patients | at time of surgery, after 7-14 days of gefitinib

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Mayer, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee